CLINICAL TRIAL: NCT00766311
Title: Aerobic and Strengthening Exercise for Acute Leukemia
Acronym: XRCISL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: XRCISL
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Hand Strength; Pliability; Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): This single-arm feasibility trial will evaluate the administration of an aggressive exercise regimen.
  Interventions: Other: Gross Motor Function; Other: Knee extension strength; Other: Hand grip strength; Other: Flexibility; Other: Ankle range of motion; Other: Aerobic capacity; Other: Body composition and vital signs

INTERVENTIONS:
Other: Gross Motor Function — The Bruinicks-Osteretsky Test of Motor Proficiency Version 2 (BOT-2) will be used to measure participants' motor function. The test is norm- referenced and designed to test motor function in children and adolescents 4 -21 years of age. The motor composite score describes overall motor abilities and is comprised of fine motor control, manual coordination, body coordination, and strength and agility. We will use the total motor composite to describe overall motor function.
Other: Knee extension strength — Maximum isometric knee extension strength will be measured with the subject seated in an adjustable straight-back chair. The pelvis will be fixed by an adjustable strap and the knee flexed to 45 degrees. The participant will exert a maximal voluntary force until their contraction is "broken."
Other: Hand grip strength — Hand grip strength in kilograms will be measured using a Jamar hand held dynamometer (Sammons Preston Rolyan, Nottinghamshire, UK). Participants will be seated with the shoulder at 0-10 degrees and the elbow in 90 degrees of flexion. The forearm will be positioned in neutral. Each participant will complete three trials, and the average used for analysis.
Other: Flexibility — Flexibility will be measured by having the participant perform the sit and reach test. A yardstick is placed on a firm flat surface and tape is placed across it at a right angle to the 15 inch mark. The participant sits with the yardstick between the legs with legs extended at right angles to the taped line on the floor. The heels of the feet touch the edge of the taped line and are 10-12 inches apart. The participant reaches forward with both hands as far as possible, keeping the hands parallel. The best value for three trials, in centimeters, at the most distant point of the fingertips is recorded.
Other: Ankle range of motion — Ankle dorsiflexion active and passive range of motion will be measured with a goniometer. The goniometer is a reliable and valid measure of active and passive range of motion if the rater uses standard procedures
Other: Aerobic capacity — Participants will complete the modified Cooper test where they walk in a corridor as fast as possible for six minutes. The distance is recorded in meters and can also be used to estimate peak V02
Other: Body composition and vital signs — Height, body mass index, waist circumference, and blood pressure will be measured.

SUMMARY:
Survivors of childhood leukemia have muscle weakness and impaired mobility (physical performance), a higher than expected frequency of obesity, and early mortality from cardiovascular disease. Treatment related neuropathy, cardiotoxicity and general cachexia may complicate physical performance and establish a pattern of sedentary behavior that may lead to a lifetime of inactivity. There is limited evidence that children being treated for leukemia benefit from home exercise programs during the maintenance phase of therapy, particularly in terms of muscle strength and range of motion. However, there are no established guidelines regarding the prescription of exercise for children diagnosed with leukemia. We propose to test the feasibility of an exercise intervention among children being treated for acute lymphoblastic leukemia (ALL) and hypothesize that children who participate in the exercise intervention will demonstrate improvements in gross motor function, strength, flexibility, and cardio respiratory fitness, and that they will have more favorable body composition when compared to the children who are assigned to the usual activity group.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the feasibility of an aerobic and strengthening exercise intervention trial among children during maintenance therapy for childhood ALL by evaluating participant accrual, participant compliance, and burden to the institutional staff.

We anticipate that key barriers exist which threaten the successful completion of an interventional trial of exercise within the ALL patient population. Approximately 2,500 to 3,500 children are diagnosed each year with ALL and similar numbers will enter the maintenance phase of therapy during a given year. About 22% of those diagnosed are between 5 and 8 years old. Thus accrual is limited by the small patient population but fortunately most patients with ALL receive their care at dedicated pediatric oncology institutions. Lack of interest or lack of understanding of the underlying problem of obesity and weakness among survivors in the ALL population may be additional barriers to accrual. In addition, families may be overwhelmed by the primary diagnosis of leukemia and feel that they are unable to take on additional challenges.

Compliance to a rigorous exercise regimen must be ascertained if demonstrable improvement in motor performance, body composition and cardiovascular disease risk profile are to occur. Key to this study is not only short-term compliance but designing an intervention that will promote and improve long-term rates of exercise. Barriers to compliance include length of time to complete the intervention, number of days the intervention must be administered, perceived benefit by the participant, difficulty of the intervention, inadequate demonstration of the intervention, poor understanding by the participant/parent of the importance of obesity and weakness among survivors of childhood ALL, and health issues in regard to the primary diagnosis of ALL.

We will open a feasibility study at 3 institutions dedicated to treatment of childhood cancer: St. Jude Children's Research Hospital, Oregon Health & Science University and Vanderbilt Ingram Cancer Center .The accrual goal of this study will be a total of 20 patients. The hypothesized outcome for this aim of the feasibility study will be an accrual rate of 50% of eligible patients at a given institution.

Motor Function The Bruinicks-Osteretsky Test of Motor Proficiency Version 2 (BOT-2) will be used to measure participants' motor function. Maximum isometric knee extension strength will be measured with a hand held myometer and hand grip strength will be measured with a hand held dynamometer. Additionally, flexibility will be measured with the sit and reach test. Ankle dorsiflexion active and passive range of motion will be measures with a goniometer. Aerobic capacity will be measured with the modified Cooper 6 minute walk test. Body composition and vital signs will also be collected.

Intervention Participants will receive counseling and written material regarding the benefits of exercise and an individualized exercise instruction session based on the results of their baseline testing and their individual preferences. Each program will include ability specific stretching/flexibility, progressive resistive strengthening, and aerobic exercise. Necessary equipment for the strengthening (weights, stretch cords, elastic bands) and aerobic components will also be provided. A videotape demonstrating each exercise in the intervention will be given to the participant and their parent."

Detailed written instructions, along with a book to log exercise, will also be provided. Stickers and small toys will be provided for the parents to give to their children for completing their exercises. Participants will receive a weekly phone call from an exercise coach, to answer questions and to progress the intervention. Participants will also receive counseling and review/progression of the exercise intervention at each usual clinic visit (approximately monthly). During the pilot study, participants will continue to receive the intervention for six months, with weekly phone calls tapering to every other week after three months. The exercise coach will be available to the participant/parent as needed via phone and/or email throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with childhood ALL when age greater than 1 and less than 10 at diagnosis, white blood cell count less than 50,000 cells/microliter and receiving continuation/maintenance therapy based on the original disease classification
* In first remission
* Maintenance phase of therapy (Eligibility extends from Day 0 of maintenance therapy up to six months prior to the completion of therapy)
* Current age 5-10 years
* Modified Lansky performance scale must score 60 or higher at time of enrollment
* Written informed consent

Exclusion Criteria:

* Lower extremity amputation or congenital deformity of lower limb
* History of pre-existing neuron-motor or neuro-developmental disorder prior to diagnosis of childhood ALL, such as mental retardation, Down syndrome, cerebral palsy, and traumatic brain injury
* Pre-existing heart or lung disease by clinical history
* Children with specific contraindications to exercise will be offered enrollment after this transient condition is resolved: severe anemia (Hemoglobin less than 8 g/dl), fever greater than 38 degrees Centigrade, platelets less than 50*109/ul, neutrophil counts less than 0.5*109/ul.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of an aerobic and strengthening exercise intervention trial among children during maintenance therapy for childhood ALL by evaluating participant accrual, participant compliance and burden to institutional staff. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (4):
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org